CLINICAL TRIAL: NCT04220619
Title: Rescue Transesophageal Echocardiography for the Guidance of Cardiopulmonary Resuscitation for In-hospital Cardiac Arrest Versus Conventional ACLS
Brief Title: RescueTEE for In-hospital Cardiac Arrest (ReTEECA Trial)
Acronym: ReTEECA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough resources to execute study
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Asad Usman, MD, MPH, Co-Primary Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 850190
Record Dates: First submitted 2019-08-27; First posted 2020-01-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Echocardiography, Transesophageal; In-hospital Cardiac Arrest; Cardiac Arrest; Cardiopulmonary Arrest With Successful Resuscitation; ACLS; Image Guided ACLS
Keywords: Cardiac Arrest; Transesophageal Echocardiography; CPR; Image Guided CPR; Conventional CPR; RescueTEE
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Convenience Sampled, Prospective Arm1: Conventional ACLS Arm2: Image Guided RescueTEE ACLS
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Conventional ACLS and Rescue TEE ALCS patients after codes will be observed for survival. Care teams will be blinded to the methodology of ACLS.
  A post-hoc analysis will also be performed for independent ECHO reads.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conventional ACLS (No Intervention): Patients who have conventional ACLS during in-hospital Cardiac arrest, they will not have RescueTEE
- RescueTEE guided ACLS (Experimental): Patients who have RescueTEE guided ACLS
  Interventions: Diagnostic Test: Tranesophageal Echocardiography

INTERVENTIONS:
Diagnostic Test: Tranesophageal Echocardiography — RescueTEE during ACLS versus Conventional ACLS
  Arms: RescueTEE guided ACLS

SUMMARY:
ReTEECA Trial. Rescue TransEsophageal Echocardiography for In-Hospital Cardiac Arrest.

This trial is aimed at studying the utility and interventional outcomes of rescue transesophageal echocardiography (RescueTEE) to aid in diagnosis, change in management, and outcomes during CPR by using a point of care RescueTEE protocol in the evaluation of in-hospital cardiac arrest (IHCA). This is an interventional prospective convenience sampled partially blinded phase II clinical trial with primary outcomes of survival to hospital discharge (SHD) with RescueTEE image guided ACLS versus conventional ACLS.

DETAILED DESCRIPTION:
This is a Phase II, single center, partially blinded, prospective, safety and efficacy pragmatic clinical trial comparing rescue transesophageal image guided ACLS versus conventional ACLS in adult patients with in-hospital cardiac arrest (IHCA). The ReTEECA Trial will use a recently published and validated focused 5-view RescueTEE protocol to evaluate patients with IHCA to obtain diagnostic and therapeutic information to aid in medical decision-making in a rapid fashion for those patients who are experiencing in-hospital arrest.1 Patients will be resuscitated with one of the following protocols:

1. Conventional ACLS with RescueTEE during IHCA. The TEE probe will be brought to the IHCA code call and placed within 10 minutes of cardiac arrest after a secured airway has been obtained. The RescueTEE team led by a physician (RescueTEE MD) and will use a predefined protocol for diagnosis and if needed intervention at the discretion of the treating physician (Code Team MD). If an intervention is performed this will be done at the discretion of the treating physician as a pragmatic and clinically evidenced intervention. The TEE probe will remain indwelling for 30 minutes or until return of spontaneous circulation (ROSC) whichever is earlier.
2. Conventional ACLS without RescueTEE during IHCA. Conventional ACLS will be driven by national American Heart Association (AHA) standardized protocols by the treating physician (Code Team MD) and code team members.

Management of the patient and ACLS will be driven pragmatically and by the local code team (Code Team MD) and not the RescueTEE team. Advice and diagnostic evidence, as able, from the RescueTEE will be provided by the RescueTEE team (RescueTEE MD). Post ROSC care will be at the discretion of the ICU team (ICU MD). The indications for using a validated published RescueTEE protocol is to study the outcome effects of an intervention that is publicly available and apply this in a real-world clinical scenario as a prospective trial.

Based on our preliminary results we hypothesize that routine use of RescueTEE guided ACLS for IHCA will expedite diagnosis, treatment, intervention, and facilitate and identify reversible causes and significantly improve survival to hospital discharge and in turn functional survival compared to standard ACLS.

Given the poor clinical outcomes of IHCA it is imperative to conduct research in this area. RescueTEE provides an avenue to help diagnose and clinically intervene on pathology during the intra-arrest period. This directly impacts the disease process, the patient, and will likely change ACLS management. There are studies that have been conducted retrospectively and prospectively that highlight the benefits of image guidance during ACLS; however, no randomized clinical trial documenting the safety and efficacy of RescueTEE has been conducted. Many institutions and hospital systems are now using RescueTEE during ACLS; however, we do not know the impact that this has had directly on survival and complications. Like many areas in medicine, a prospective clinical trial can help elucidate the direct patient benefits in terms of survival. This will offer future researchers a platform to conduct further studies on image guidance during ACLS. A prospective clinical trial is necessary to transform national guidelines and help guide evidence-based practice throughout the country.

ReTEECA Trial Hypothesis: Based on our preliminary results we hypothesize that routine use of RescueTEE guided ACLS for IHCA will expedite diagnosis, treatment, intervention, and facilitate and identify reversible causes and significantly improve survival to hospital discharge and in turn functional survival compared to standard ACLS.

ReTEECA Trial: We propose a Phase II, single center, partially blinded, intention to treat, safety and efficacy clinical trial to assess the results of routine RescueTEE guided ACLS for IHCA compared with standard ACLS. The Hospital of the University of Pennsylvania and the Department of Anesthesiology and Critical Care has the patient population, experience, expertise, and infrastructure to execute the proposed study.

Specific Aims: The goal of the study will be to use intra-arrest RescueTEE diagnostic imaging to guide the code leader in clinical management and decision-making and to therefore decrease IHCA mortality rates. Additionally, we will assess if RescueTEE guidance of intra-arrest therapies or interventions can significantly improve functionally favorable outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients greater than 18 years of age;
* Intubated or permanent tracheostomy in situ;
* Experiencing extreme hemodynamic instability, cardiac arrest, or respiratory arrest and TTE is difficult or contraindicated
* Rapid response, Code calls, ECMO stat evaluation
* In-patients

Exclusion Criteria:

* Unsecured airway
* On-going aspiration
* History of tracheoesophageal injury
* History of tracheoesophageal fistula
* Esophagectomy
* Active upper GI bleeding
* Esophageal varices
* Ongoing hemoptysis
* Technically challenging TEE placement due to location of code - Small room, intrusive to the code team, airway trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 3 months
  Survival to hospital discharge (SHD) - Survival is the most widely accepted endpoint in CPR and CA trials. Our trial is designed to evaluate the effect of imaging and RescueTEE guided ACLS in order to facilitate survival.

SECONDARY OUTCOMES:
Number of patients surviving to End of ACLS | 1 hour
  Count of patients surviving to End of Code
Number of patients surviving to ICU discharge | Variable
  Count of patients surviving to ICU discharge
Number of patients surviving to 30 days | 30 days
  30 days survival for image guided RescueTEE ACLS versus conventional ACLS
Neurologically Intact Survival at 3 months | 3 months
  Neurologically intact survival based on modified Rankin's Score at 3 month
Neurologically Intact Survival at 6 months | 6 months
  Neurologically intact survival based on modified Rankin's Score at 6 month

OTHER OUTCOMES:
Optimal Hand Positioning | 1 hour
  Comparing baseline hand positioning versus RescueTEE guided hand positioning during cardiac arrest.
  The echocardiographer will use RescueTEE to optimize hand positioning during cardiac arrest. This information will be documented before and after changing hand positioning to determine if there was a resultant change in ROSC. We will assess if optimization of hand positioning over the area of maximal impulse (AMI) during chest compressions based on TEE results in increased likelihood of ROSC
Feasibility and safety of TEE probe insertion during CPR | 10 minutes
  To calculate the failure rates, feasibility, and technical issues in placing TEE probes during ACLS. This will be determined by asking code leaders to fill up a follow up form to reflect a qualitative feedback to see if TEE was useful in a subjective manner. We will also calculate the time from code to TEE probe insertion and also the time for total examination. Data will be collected on the technical challenges encountered with probe placement. Post-event images will be reviewed and quality will be assessed in terms of clarity, motion artifact, and reproducibility.
Image quality | 1 hour
  To document the imaging quality and diagnostic capabilities of RescueTEE during ACLS. A blinded reviewer will perform QI on the image quality. This will be a descriptive statistic looking at contrast, gain both lateral and medial gain, overgain, image depth, focus length. Numerical outcomes of which views were obtained from the 5 selected views. These will be reported as standard echocardiography image quality assessments are done for clinical practice.
Diagnoses of pathology in image guided ACLS | 1 hour
  Descriptive statistics: To document the range of diagnoses RescueTEE can provide during CPR in the management of in-hospital arrest or critical hemodynamic instability. The RescueTEE form competed by the echocardiographer lists several diagnoses including the following: cardiac tamponade, LV thrombus, RV thrombus, fine VF, Pulseless rhythm with echocardiographic evidence of motion (PREM) versus Pulseless rhythm with echocardiographic evidence of standstill (PRES), myocardial infarction, aortic dissection, severe hypovolemia, severe global LV dysfunction, severe global RV dysfunction, and LV free wall rupture.
Interventional and therapeutic support during image guided ACLS | 1 hour
  Descriptive statistics: To document and classify the role that RescueTEE can provide which leads to therapeutic guidance or intervention for the code leader during arrest situations. Information regarding the interventions will include TEE driven medication administration or procedural management. This will also be recorded as a categorical variable as; fluid given, blood given, epinephrine given, shock advised for pulseless rhythm with echocardiographic evidence of motion (PREM), calcium given, pericardiocentesis performed, ECMO cannulation completed, thrombolytics administered, or chest compressions hand positioning changed, or chest compressions terminated.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Gutsche, MD, Principal Investigator — University of Pennsylvania, Department of Anesthesiology and Critical Care; Asad A Usman, MD, MPH, Principal Investigator — University of Pennsylvania, Department of Anesthesiology and Critical Care

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaspari R, Weekes A, Adhikari S, Noble V, Nomura JT, Theodoro D, Woo M, Atkinson P, Blehar D, Brown S, Caffery T, Douglass E, Fraser J, Haines C, Lam S, Lanspa M, Lewis M, Liebmann O, Limkakeng A, Lopez F, Platz E, Mendoza M, Minnigan H, Moore C, Novik J, Rang L, Scruggs W, Raio C. A retrospective study of pulseless electrical activity, bedside ultrasound identifies interventions during resuscitation associated with improved survival to hospital admission. A REASON Study. Resuscitation. 2017 Nov;120:103-107. doi: 10.1016/j.resuscitation.2017.09.008. Epub 2017 Sep 13. PMID 28916478
- [Background] Markin NW, Gmelch BS, Griffee MJ, Holmberg TJ, Morgan DE, Zimmerman JM. A review of 364 perioperative rescue echocardiograms: findings of an anesthesiologist-staffed perioperative echocardiography service. J Cardiothorac Vasc Anesth. 2015 Feb;29(1):82-8. doi: 10.1053/j.jvca.2014.07.004. Epub 2014 Nov 7. PMID 25440641
- [Background] Min JK, Spencer KT, Furlong KT, DeCara JM, Sugeng L, Ward RP, Lang RM. Clinical features of complications from transesophageal echocardiography: a single-center case series of 10,000 consecutive examinations. J Am Soc Echocardiogr. 2005 Sep;18(9):925-9. doi: 10.1016/j.echo.2005.01.034. PMID 16153515
- [Background] Staudt GE, Shelton K. Development of a Rescue Echocardiography Protocol for Noncardiac Surgery Patients. Anesth Analg. 2019 Aug;129(2):e37-e40. doi: 10.1213/ANE.0000000000003569. PMID 29916865
- [Background] Long B, Alerhand S, Maliel K, Koyfman A. Echocardiography in cardiac arrest: An emergency medicine review. Am J Emerg Med. 2018 Mar;36(3):488-493. doi: 10.1016/j.ajem.2017.12.031. Epub 2017 Dec 16. PMID 29269162
- [Background] Gaspari R, Weekes A, Adhikari S, Noble VE, Nomura JT, Theodoro D, Woo M, Atkinson P, Blehar D, Brown SM, Caffery T, Douglass E, Fraser J, Haines C, Lam S, Lanspa M, Lewis M, Liebmann O, Limkakeng A, Lopez F, Platz E, Mendoza M, Minnigan H, Moore C, Novik J, Rang L, Scruggs W, Raio C. Emergency department point-of-care ultrasound in out-of-hospital and in-ED cardiac arrest. Resuscitation. 2016 Dec;109:33-39. doi: 10.1016/j.resuscitation.2016.09.018. Epub 2016 Sep 28. PMID 27693280
- [Background] Arntfield R, Lau V, Landry Y, Priestap F, Ball I. Impact of Critical Care Transesophageal Echocardiography in Medical-Surgical ICU Patients: Characteristics and Results From 274 Consecutive Examinations. J Intensive Care Med. 2020 Sep;35(9):896-902. doi: 10.1177/0885066618797271. Epub 2018 Sep 6. PMID 30189783
- [Background] Daniel WG, Erbel R, Kasper W, Visser CA, Engberding R, Sutherland GR, Grube E, Hanrath P, Maisch B, Dennig K, et al. Safety of transesophageal echocardiography. A multicenter survey of 10,419 examinations. Circulation. 1991 Mar;83(3):817-21. doi: 10.1161/01.cir.83.3.817. PMID 1999032
- [Background] Fair J, Mallin M, Mallemat H, Zimmerman J, Arntfield R, Kessler R, Bailitz J, Blaivas M. Transesophageal Echocardiography: Guidelines for Point-of-Care Applications in Cardiac Arrest Resuscitation. Ann Emerg Med. 2018 Feb;71(2):201-207. doi: 10.1016/j.annemergmed.2017.09.003. Epub 2017 Nov 6. PMID 29107407
- [Background] Shillcutt SK, Markin NW, Montzingo CR, Brakke TR. Use of rapid "rescue" perioperative echocardiography to improve outcomes after hemodynamic instability in noncardiac surgical patients. J Cardiothorac Vasc Anesth. 2012 Jun;26(3):362-70. doi: 10.1053/j.jvca.2011.09.029. Epub 2012 Jan 4. PMID 22226417
- [Background] Teran F, Dean AJ, Centeno C, Panebianco NL, Zeidan AJ, Chan W, Abella BS. Evaluation of out-of-hospital cardiac arrest using transesophageal echocardiography in the emergency department. Resuscitation. 2019 Apr;137:140-147. doi: 10.1016/j.resuscitation.2019.02.013. Epub 2019 Feb 16. PMID 30779977